CLINICAL TRIAL: NCT02125786
Title: A Phase II Trial of Surgery and Fractionated Re-Irradiation for Recurrent Ependymoma
Brief Title: A Trial of Surgery and Fractionated Re-Irradiation for Recurrent Ependymoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RERTEP; NCI-2014-00906 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Results first posted 2024-11-12 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Ependymoma
MeSH Terms: conditions — Ependymoma | interventions — Radiation; Craniospinal Irradiation; Surgical Procedures, Operative; Metastasectomy; Fluorodeoxyglucose F18; Contrast Media; Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Stratum 1: Local Failure (Experimental): Participants exhibit an initial pattern of failure that is local (disease confined to primary site). Treatment is surgery and a second course of focal irradiation. The total dose for the second course of irradiation will be 54Gy.
  Participants may receive one or both: Photon therapy or proton therapy.
  Participants receive ^1^8F-fluorodeoxyglucose and ^1^1C-methionine to aid in tumor visualization.
  Interventions: Radiation: Irradiation; Procedure: Surgery; Drug: ^1^8F-Fluorodeoxyglucose; Drug: ^1^1C-methionine; Device: Photon therapy; Device: Proton therapy
- Stratum 2: Metastatic Failure (Experimental): Participants exhibit an initial pattern of failure that is metastatic (neuraxis metastatic disease without equivocal evidence of local failure). Treatment is surgery and craniospinal irradiation. Craniospinal irradiation (36-39.6Gy) will include focal boost treatment of metastatic sites (54-59.4Gy) depending on location, extent of resection and target volume.
  Participants may receive one or both: Photon therapy or proton therapy.
  Participants receive ^1^8F-fluorodeoxyglucose and ^1^1C-methionine to aid in tumor visualization.
  Interventions: Radiation: Irradiation; Procedure: Surgery; Drug: ^1^8F-Fluorodeoxyglucose; Drug: ^1^1C-methionine; Device: Photon therapy; Device: Proton therapy
- Stratum 3: Local and Metastatic Failure (Experimental): Participants exhibit an initial pattern of failure that is both local and metastatic (neuraxis metastatic disease with equivocal evidence of local failure). Treatment is surgery and craniospinal irradiation.
  Participants may receive one or both: Photon therapy or proton therapy.
  Participants receive ^1^8F-fluorodeoxyglucose and ^1^1C-methionine to aid in tumor visualization.
  Interventions: Radiation: Irradiation; Procedure: Surgery; Drug: ^1^8F-Fluorodeoxyglucose; Drug: ^1^1C-methionine; Device: Photon therapy; Device: Proton therapy
- Stratum 4: Local Failure (Experimental): Local Failure Participants exhibit an initial pattern of failure that is local (disease confined to primary site). Age is >36 months at time of enrollment to <21 years. Tumor shows presence of 1q gain. Treatment is optional craniospinal irradiation.
  Participants may receive one or both: Photon therapy or proton therapy.
  Participants receive ^1^8F-fluorodeoxyglucose and ^1^1C-methionine to aid in tumor visualization.
  Interventions: Radiation: Irradiation; Procedure: Surgery; Drug: ^1^8F-Fluorodeoxyglucose; Drug: ^1^1C-methionine; Device: Photon therapy; Device: Proton therapy

INTERVENTIONS:
Radiation: Irradiation — Radiation therapy on this protocol will be based on extent of disease, extent of resection and location. The allowed treatment modalities include conformal or intensity-modulated radiation therapy using photons or proton therapy using double-scattering or spot-scanning methods. The general goal is to initiate radiation therapy within 12 weeks of last surgery performed at the time of recurrence.
  Other Names: Focal irradiation; Craniospinal irradiation
Procedure: Surgery — When applicable, surgery will be used to remove metastases. The goal of surgery is to achieve gross total resection of all imaging visible residual tumor.
  Other Names: Metastasectomy
Drug: ^1^8F-Fluorodeoxyglucose — This is a contrast media that will be given intravenously to aid in tumor visualization.
  Other Names: 18F-FDG; Contrast Media
Drug: ^1^1C-methionine — This is a contrast media that will be given intravenously to aid in tumor visualization.
  Other Names: Contrast Media
Device: Photon therapy — Participants will receive one or both: Photon or proton therapy.
  Other Names: Photon linear accelerator
Device: Proton therapy — Participants will receive one or both: Photon or proton therapy.
  Other Names: Proton synchroton

SUMMARY:
The primary purpose of this study is to investigate whether surgery and re-irradiation will help treat ependymoma that has come back after initial treatment. The combined doses of the first and second courses of radiation are higher than what is usual standard of care. The investigators will study the effects and side effects of surgery and re-irradiation. They will also evaluate and study tumor tissue and blood to learn more about the tumor and how it does or does not respond to treatments and will use magnetic resonance imaging (MRI) and positron emission tomography (PET) scans to see if they can predict tumor response and tumor recurrence.

Participants will be followed for up to 5 years following enrollment. Evaluations during radiation therapy will be done weekly while receiving therapy for up to 7 weeks. Other evaluations will be done at enrollment, every 4 months from enrollment through 3 years, and every 6 months during the 4th and 5th year.

DETAILED DESCRIPTION:
Stratification for treatment will be determined when radiation therapy planning is initiated. Patients will be stratified for outcome according to diagnosis and prior therapy.

* Stratum 1 (initial pattern of failure is local); disease confined to primary site; age >12 months at time of enrollment to < 21 years. Treatment: focal irradiation.
* Stratum 2 (initial pattern of failure is metastatic); neuraxis metastatic disease without equivocal evidence of local failure; age > 36 months at time of enrollment to < 21 years. Treatment: craniospinal irradiation.
* Stratum 3 (Initial pattern of failure is both local and metastatic): neuraxis metastatic disease with unequivocal evidence of local failure; age > 36 months at time of enrollment to < 21 years. Treatment: craniospinal irradiation.
* Stratum 4 (initial pattern of failure is local): disease confined to primary site, age >36 months at time of enrollment to <21 years; tumor shows presence of 1g gain. Treatment: craniospinal irradiation (optional).

PRIMARY OBJECTIVE:

* To prospectively estimate the progression-free and overall survival distributions for children and young adults with recurrent ependymoma treated with a second course of irradiation while monitoring for excessive central nervous system necrosis.

SECONDARY OBJECTIVES:

* To explore potential associations of clinical and treatment factors with the incidence and severity of neurological, endocrine and cognitive deficits in children and young adults with ependymoma treated with a second course of irradiation.
* Using specific measures of sleep quality, excessive daytime sleepiness, daytime activity, fatigue, symptom distress, and quality of life, explore associations of sleep, fatigue and quality of life with other measures of CNS effects, clinical and treatment factors in children and young adults with ependymoma treated with a second course of irradiation.
* To evaluate and explore differences in physical performance and movement in children and young adults with ependymoma treated with a second course of irradiation.
* Estimate and compare the response of residual tumor and the incidence and severity of structural, physiological, and vascular effects of normal brain in children and young adults with ependymoma after treatment with a second course of irradiation using specific methods of diffusion, contrast-enhancement, magnetization transfer, vascular and functional neuroimaging, and explore the association between these and other measures of CNS effects and clinical and treatment factors. Determine the time course of gray matter and white matter tract injury and recovery post irradiation and the association between imaging metrics derived from serial quantitative neural imaging and radiation dosimetry as well as neuro-cognitive outcomes.

Other Pre-Specified (Exploratory) Objectives:

* Estimate the avidity of ependymoma to 18F-fluorodeoxyglucose (FDG) and 11C-methionine positron emission tomography (IND # 104987) prior to radiation therapy and correlate change in avidity 12, 24 and 36 months after a second course of irradiation with tumor progression.
* Measure growth factor and cytokine responses in children and young adults with ependymoma after treatment with a second course of irradiation, and explore associations between these and other measures of CNS effects and clinical and treatment factors. Descriptively compare findings for patients treated with an initial course of irradiation.
* To conduct a variety of exploratory molecular analyses on tumor samples (and blood where a germline control is required), including but not limited to broad (genome-wide / array-based) or focused (gene-specific) analyses at the DNA, RNA, or protein level and next generation (whole genome, exome, transcriptome) sequencing in an effort to improve the investigators understanding of ependymoma biology, and to explore associations between molecular findings and treatment response and various side effects including vasculopathy, hearing loss, cognitive deficits, and growth hormone deficiency and other measures as appropriate.
* To explore the association of chemotherapy given prior to re-irradiation with progression-free survival and overall survival distributions
* To compare the progression-free and overall survival distributions for children (age >3 years) and young adults with recurrent ependymoma and 1g gain treated with a second course of irradiation (focal or craniospinal) while monitoring for excessive central nervous system necrosis.

ELIGIBILITY:
Inclusion Criteria:

* Progressive intracranial ependymoma after prior focal irradiation
* Patients aged 1-21 years at the time of enrollment
* Adequate performance status (ECOG < 3) and research participant does not require mechanical ventilation
* Interval from start of initial radiation therapy to enrollment > 9 months

Exclusion Criteria:

* Prior craniospinal irradiation
* Pregnant women are excluded from enrollment on this study because radiation therapy is an agent with the potential for teratogenic or abortifacient effects
* Any patient with both metastatic ependymoma and age < 3 years at the time of enrollment

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2014-05-07 (Actual); Primary Completion 2023-05 (Actual); Study Completion 2028-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Merchant, DO, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 enrollments occurred on 68 participants between from April 21, 2014 and June 30, 2020.
Pre-assignment Details: Of 70 enrollments, 3 were found to be ineligible and removed; 3 withdrew before reirradiation to seek other treatment. One participant who was initially ineligible was later found to be eligible and re-enrolled, and a participant who had previously withdrawn to seek other treatment options decided to pursue reirradiation and re-enrolled. The 2 screen failures St. Jude pathology did not result ependymoma diagnosis after consent as expected. Sixty-four (64) completed reirradiation treatment.
Groups:
- Reirradiation: Children and young adults with Recurrent Ependymoma undergoing reirradiation
Period: Overall Study
Arm/Group | Reirradiation
Started | 68
Completed | 9
Not Completed | 59
Not completed — Still in Follow-up | 3
Not completed — Screen Failure | 2
Not completed — Withdrawal by Family before Start of RT | 2
Not completed — Progressive Disease | 44
Not completed — Death | 8

BASELINE CHARACTERISTICS:
Population: Children and young adults with Recurrent Ependymoma undergoing reirradiation.
Arm/Group | Reirradiation
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.95 (5.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 51
  More than one race | 2
  Unknown or Not Reported | 0
Treatment Stratum [Count of Participants; unit: Participants]
  Stratum 1(Initial pattern of failure is local) Treatment: Focal Irradiation | 25
  Stratum 2 (Initial pattern of failure is metastatic) Treatment: CSI | 16
  Stratum 3 (Initial pattern of failure is local and metastatic) Treatment: CSI | 15
  Stratum 4 (Initial pattern of failure is local) Treatment: CSI (optional-presence of 1q gain & >3yo) | 8

OUTCOME MEASURES:

1. Primary Outcome: 3-year Progression-free Survival Rate
Description: To prospectively estimate the progression-free distribution for children and young adults with recurrent ependymoma treated with a second course of irradiation.
Time Frame: 2 years follow-up after initiation of radiation therapy for the last patient enrolled
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Reirradiation
Number analyzed (Participants) | 64
percentage of participants | 21.88 [12.73 to 32.61]

2. Primary Outcome: 3-year Overall Survival Rate
Description: OS was calculated from the date of initial radiation therapy to date of death or date of last contact for the patients who were treated with RT. The event of interest was death.
Time Frame: 2 years follow-up after initiation of radiation therapy for the last patient enrolled
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Reirradiation
Number analyzed (Participants) | 64
percentage of participants | 60.33 [47.14 to 71.20]

3. Secondary Outcome: Incidence Rate of Neurological Deficits
Description: Evaluation will be in children and young adults with ependymoma treated with a second course of irradiation.
  Outcomes will be reported by p-values.
Time Frame: Through 5 years after initiation of second course of irradiation
Reporting Status: Not Posted

4. Secondary Outcome: Incidence Rate of Ophthalmological Deficits
Description: Evaluation will be in children and young adults with ependymoma treated with a second course of irradiation.
  Outcome will be reported with p values.
Time Frame: Through 5 years after initiation of second course of irradiation
Reporting Status: Not Posted

5. Secondary Outcome: Incidence Rate of Audiological Deficits
Description: Evaluation will be in children and young adults with ependymoma treated with a second course of irradiation.
  Outcome will be reported with p-values.
Time Frame: Through 5 years after initiation of second course of irradiation
Reporting Status: Not Posted

6. Secondary Outcome: Incidence Rate of Endocrine Deficits
Description: as for outcome 5
Time Frame: Through 5 years after initiation of second course of irradiation
Reporting Status: Not Posted

7. Secondary Outcome: Number of Neurocognitive Deficits
Time Frame: Through 5 years after initiation of second course of irradiation
Reporting Status: Not Posted

8. Secondary Outcome: Mean Change in Quality of Life by Treatment Arm
Description: Baseline is defined as day 1 of radiation therapy.
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

9. Secondary Outcome: Mean Change in Measured Task Sets
Description: Baseline is defined as day 1 of radiation therapy.
  Measured task sets: BOT2 (4-21 years old) and PPT (≥22 years old).
  * BOT2 outcome: total motor composite, a standardized score range from 20 to 80, with a mean of 50 and a standard deviation of 10.
  * PPT (7-item questionnaire) outcome: a score range from 0 to 28. The normative data is available from the human performance lab.
  The above scores will be standardized into z-scores/T-scores for data analysis based on normative data.
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

10. Secondary Outcome: Mean Change in Physical Function
Description: Baseline is defined as day 1 of radiation therapy.
  Self-reported instruments (PROMIS): Three questionnaires.
  * Pediatric Physical Function - Mobility - SF1: 8-item questionnaire with the score range from 0 to 32.
  * Pediatric Physical Function - Upper Extremity - SF1: same as above.
  * Physical Function - SF1: 10-item questionnaire with the score range from 0 to 50.
  The above scores will be standardized into z-scores/T-scores for data analysis based on normative data
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

11. Secondary Outcome: Mean Change in Body Mass Index (kg/m2)
Description: Baseline is defined as day 1 of radiation therapy
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

12. Secondary Outcome: Mean Change in Waist/Hip Ratio (cm/cm)
Description: Baseline is defined as day 1 of radiation therapy.
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

13. Secondary Outcome: Mean Change in Ankle Dorsiflexion
Description: Baseline is defined as day 1 of radiation therapy.
  Ankle dorsiflexion active and passive range of motion: measured by goniometer, and recorded as an angle (degree).
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

14. Secondary Outcome: Mean Change in Overall Flexibility in cm
Description: Baseline is defined as day 1 of radiation therapy.
  Overall flexibility: measured by sit and reach test, and recorded as a length (cm).
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

15. Secondary Outcome: Proportion Change in Balance
Description: Baseline is defined as day 1 of radiation therapy.
  Balance measured by Measured by sensory organization test (SOT), and the result from the test is the equilibrium score, a percentage range from 0% to 100%, with the higher percentage, the better balance. The outcome is a binary variable with a cutoff score of < 70% indicates future risk for a fall.
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

16. Secondary Outcome: Mean Change in Fine Motor Coordination
Description: Baseline is defined as day 1 of radiation therapy.
  Fine motor coordination (finger and hand coordination). Measured by Composite Cerebellar Functional Severity Score (CCFS), and the outcome is an age-adjusted z-score and log transformed.
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

17. Secondary Outcome: Mean Change in Overall Coordination
Description: Baseline is defined as day 1 of radiation therapy.
  Overall coordination measured by brief ataxia rating scale (five-item questionnaire). The outcome is a total scale range from 0 to 22.
Time Frame: Fine motor coordination (finger and hand coordination).
Reporting Status: Not Posted

18. Secondary Outcome: Mean Change of Lower Extremity Strength and Power
Description: Baseline is defined as day 1 of radiation therapy.
  Lower extremity strength measured by BiodexIII. The outcomes are peak torque value/body weight ratios at different speeds of motion.
  The scores will be standardized into z-scores for data analysis based on normative data.
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

19. Secondary Outcome: Mean Change in Hand Grip Strength
Description: Baseline is defined as day 1 of radiation therapy.
  Hand grip strength is measured by a Jamar hand held dynamometer and recorded in kilograms (kg).
  The scores will be standardized into z-scores for data analysis based on normative data.
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

20. Secondary Outcome: Mean Change in Resting Energy Expenditure
Description: Baseline is defined as day 1 of radiation therapy.
  Resting energy expenditure is measured with indirect calorimetry after an overnight fast and recorded as REE (kcal/day).
  The scores will be standardized into z-scores for data analysis based on normative data.
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

21. Secondary Outcome: Mean Change in Cardiopulmonary Exercise Test (CPET)
Description: Baseline is defined as day 1 of radiation therapy.
  Cardiopulmonary exercise test (CPET) will be completed on a treadmill using the Balke protocol or cycle ergometer using an incremental ramping protocol. The outcome is recorded as VO2max (ml/kg/min).
  The scores will be standardized into z-scores for data analysis based on normative data.
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

22. Secondary Outcome: Longitudinal Change of Size (or Extent if Leptomeningeal Dissemination) of Residual Tumor
Description: Baseline is defined as the last MRI prior to initiation of radiation therapy.
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

23. Secondary Outcome: Longitudinal Change of Incidence and Severity of Structural Effects of Normal Brain
Description: Baseline is defined as the last MRI prior to initiation of radiation therapy.
Time Frame: Baseline through 5 years after initiation of radiation therapy
Reporting Status: Not Posted

24. Secondary Outcome: Longitudinal Change in Gray and White Matter Tissues
Description: This outcome will be evaluated by neuroimaging. Baseline is defined as day 1 of radiation therapy.
Time Frame: Baseline to recovery of gray and white matter tract injury, up to a maximum of 5 years
Reporting Status: Not Posted

25. Secondary Outcome: Longitudinal Change of Individual Variation and Risk Factors in Gray and White Matter Tissues
Description: Baseline is defined as day 1 of radiation therapy.
Time Frame: Baseline to recovery of gray and white matter tract injury, up to a maximum of 5 years
Reporting Status: Not Posted

26. Secondary Outcome: Change Over Time in Imaging Metrics
Description: Baseline is defined as day 1 of radiation therapy.
Time Frame: Baseline to recovery of gray and white matter tract injury, up to a maximum of 5 years
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Avidity of Ependymoma to 18F-fluorodeoxyglucose and 11C-methionine PET Prior to Radiation Therapy
Description: Baseline is the last FDG-PET and MET-PET prior to initiation of radiation therapy.
Time Frame: Baseline
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Longitudinal Change of Avidity of Ependymoma to 18F-fluorodeoxyglucose and 11C-methionine PET Prior to Radiation Therapy
Description: Correlation of avidity of ependymoma to 18F-fluorodeoxyglucose and 11C-methionine PET prior to radiation therapy with progression-free survival will be reported
Time Frame: 12, 24 and 36 months after second course of irradiation
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Longitudinal Change of Necrosis Measured With MET/FDG and Necrosis Measured With MRI
Description: Association between necrosis measured with MET/FDG vs. MRI Baseline is defined as day 1 of radiation therapy (RT).
Time Frame: Baseline, and at 12, 24 and 36 month
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Mean Change Over Time in Cytokine Levels
Description: Baseline is defined as day 1 of radiation therapy.
Time Frame: Baseline through 5 years after radiation therapy
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Genetic Variations in Germline
Description: Evaluate will be of genetic variations in germline associated with treatment response and side effects. P-values will be reported.
  Baseline is defined as day 1 of radiation therapy.
Time Frame: Baseline
Reporting Status: Not Posted

32. Other Pre Specified Outcome: 3-year Progression-free Survival (PFS) Rates by Chemotherapy Groups
Time Frame: 2 years after initiation of irradiation for the last patient enrolled
Reporting Status: Not Posted

33. Other Pre Specified Outcome: 3 Year Overall Survival (OS) Rates by Chemotherapy Groups
Time Frame: 2 years after initiation of irradiation for the last patient enrolled
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 11C-Methionine-Related Adverse Events: From time of injection through one hour post injection of 11C-methionine. Radiation-Related Adverse Events: From initiation of radiation therapy through study completion, an average of 2 years.
Description: All-cause mortality was assessed in eligible participants who received radiation therapy. Adverse events were assessed in eligible participants with adverse event data who received radiation therapy.
Arm/Group | Reirradiation
All-Cause Mortality (participants affected / at risk) | 8/64
Serious Adverse Events (participants affected / at risk) | 2/64
Other Adverse Events (participants affected / at risk) | 30/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reirradiation (N=64)
Gastric Hemorrhage (Gastrointestinal disorders) | 1 (1) — Unrelated to radiation therapy, resulted in patient's death.
Death NOS (General disorders) | 1 (1) — Unrelated to radiation therapy, pre-existing swallowing issues developed post-operatively prior to radiation therapy; cause of death unknown as autopsy not performed.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reirradiation (N=64)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) — Associated with administration of 11C-Methionine, observed post-11C-Methionine PET scan, not radiation-related.
Sinus tachycardia (Cardiac disorders) | 3 (3) — Associated with administration of 11C-Methionine, observed post-11C-Methionine PET scan, not radiation-related.
Other-Pseudomeningocele (General disorders) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Central nervous system necrosis (Nervous system disorders) | 15 (15)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) — New diagnosis/onset of seizures.
Other - Bradypnea (Respiratory, thoracic and mediastinal disorders) | 7 (9) — Associated with administration of 11C-Methionine, observed post-11C-Methionine PET scan, not radiation-related.
Other - Tachypnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) — Associated with administration of 11C-Methionine, observed post-11C-Methionine PET scan, not radiation-related.
Hypertension (Vascular disorders) | 2 (2) — Associated with administration of 11C-Methionine, observed post-11C-Methionine PET scan, not radiation-related.
Hypotension (Vascular disorders) | 1 (1) — Associated with administration of 11C-Methionine, observed post-11C-Methionine PET scan, not radiation-related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT02125786/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT02125786/ICF_001.pdf